CLINICAL TRIAL: NCT00006206
Title: COMBINE: Effect of Combined Pharmacotherapies and Behavioral Interventions
Brief Title: COMBINE (Acamprosate/Naltrexone)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Lipha Pharmaceuticals (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAAComb; U10AA011721 (NIH); U10AA011783 (NIH); U10AA011715 (NIH); U10AA011799 (NIH); U10AA011773 (NIH); U10AA011776 (NIH); U10AA011777 (NIH); U10AA011727 (NIH); U10AA011716 (NIH); U10AA011787 (NIH); U10AA011768 (NIH); U10AA011756 (NIH); NCT00000453 (obsolete NCT alias)
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2010-05-03 (Estimated); Status verified 2007-11

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Acamprosate

INTERVENTIONS:
Drug: naltrexone (Revia)
Drug: acamprosate (Campral)

SUMMARY:
Combine is a multicenter, randomized clinical trial that will evaluate combinations of three interventions for treating alcohol dependence. The goal is to determine whether improvement in treatment outcomes can be achieved by various combinations of drug and behavioral interventions. Two of the interventions will consist of pharmacological treatment with naltrexone (Revia) or acamprosate (Campral). The third intervention is a multicomponent behavioral therapy including such components as motivational enhancement therapy, cognitive behavioral therapy, and referral to self-help groups, including AA. All three interventions will include a component supporting compliance to medications and reduction in drinking.

ELIGIBILITY:
Inclusion criteria

The following inclusion criteria are to be met:

1. Male and female outpatients > 18 years of age.
2. Participants will have a current DSM-IV diagnosis of alcohol dependence.
3. Participants will have signed a witnessed informed consent.
4. Participants must have been drinking a minimum of > 14 drinks (females) or > 21 drinks (males) on average per week over a consecutive 30-day period in the 90-day period prior to initiation of abstinence, and have two or more days of heavy drinking (defined as 4 drinks for females and 5 drinks for males) in the 90-day period prior to initiation of abstinence.
5. Participants must have had a minimum of 4 consecutive days (96 hours) of abstinence and have a CIWA < 8 prior to randomization.
6. Participants can be abstinent for a maximum of 21 days prior to randomization.
7. Participants will have no more than 21 consecutive days of planned absence during the 16 week active treatment period.
8. Participants who are able to identify at least one "locator" person to assist in tracking the participant for follow-up assessment.
9. Participants who are able to speak and understand English.

Exclusion criteria

The following exclusion criteria rule out participants:

1. Participants who meet current DSM-IV criteria for bipolar disorder, schizophrenia, bulimia/anorexia, dementia, or a psychological disorder requiring medication.
2. Participants requiring concomitant therapy with any medications that pose safety issues (see Appendix B).
3. Participants with a current diagnosis of dependence on any drug except for nicotine, cannabis, and alcohol, or habitual caffeine use. If there is a positive urine screen the participant can be retested after the (metabolic) interval appropriate to that drug. If the second urine drug screen is positive the person is excluded.
4. Participants who meet DSM-IV criteria for opiate dependence or abuse within the past 6 months, chronic treatment with any opiate-containing medications during the previous month, or urine positive for opioids.
5. Participants who have significant medical disorders that will increase the potential risk of study treatment or interfere with study participation, and participants with sensitivity to study medications or related drugs as evidenced by adverse drug experience, especially with opiate-containing analgesics, opioid antagonists, or acamprosate.
6. Participants with abnormal AST or ALT (more than 3 times the upper limit of the normal range(ULN)) or elevated bilirubin (more than 10% above the ULN). Tests may be repeated if initial results are out of range.
7. Participants who are pregnant or nursing infant(s), and women of childbearing potential not using a contraceptive method judged by the investigator to be effective.
8. Participants who intend to engage in additional formal treatment for alcohol-related problems, or who intend to continue in current treatment for alcohol-related problems during the active treatment period. Self-help treatments are not considered formal treatment.
9. Participants who have had more than seven days of inpatient treatment for substance use disorders in the 30 days previous to randomization.
10. Participants who have prior use of study medication(s) in the last 30 days.

Any question concerning the interpretation of or application of the inclusion/exclusion criteria will be referred to the medical expert at the Coordinating Center. If he is unavailable, the question will be referred to the Chairperson of the Treatment Subcommittee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1375
Dates: Start 1997-08; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent
Time to relapse to heavy drinking

SECONDARY OUTCOMES:
measures of drinking outcomes ((duration of abstinence, measures of frequency and intensity, et al.)
psychological assessments
quality of life
measures of adverse experiences

CONTACTS AND LOCATIONS:
Overall Officials: Ray Anton, M.D., Study Chair — Medical University of South Carolina
Locations (12):
- United States (12):
  - Substance Abuse Treatment Unit, Yale University, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Harvard University/McLean Hospital, Belmont, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Center on Alcoholism, Substance Abuse and Addiction, University of New Mexico, Albuquerque, New Mexico
  - Treatment and Research Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Roger Williams Medical Center , Brown University, Providence, Rhode Island
  - Center for Alcohol Programs, Medical University of South Carolina, Charleston, South Carolina
  - Southwest Texas Addiction Research and Technology Center, University of Texas Health Science Center, San Antonio, Texas
  - Addictions Treatment Center, University of Washington, Seattle, Washington
  - University of Wisconsin-Milwaukee, Milwaukee, Wisconsin

REFERENCES:
- [Background] Johnson BA, O'Malley SS, Ciraulo DA, Roache JD, Chambers RA, Sarid-Segal O, Couper D. Dose-ranging kinetics and behavioral pharmacology of naltrexone and acamprosate, both alone and combined, in alcohol-dependent subjects. J Clin Psychopharmacol. 2003 Jun;23(3):281-93. doi: 10.1097/01.jcp.0000084029.22282.bb. PMID 12826990
- [Background] COMBINE Study Research Group. Testing combined pharmacotherapies and behavioral interventions for alcohol dependence (the COMBINE study): a pilot feasibility study. Alcohol Clin Exp Res. 2003 Jul;27(7):1123-31. doi: 10.1097/01.ALC.0000078020.92938.0B. PMID 12878918
- [Background] COMBINE Study Research Group. Testing combined pharmacotherapies and behavioral interventions in alcohol dependence: rationale and methods. Alcohol Clin Exp Res. 2003 Jul;27(7):1107-22. doi: 10.1097/00000374-200307000-00011. PMID 12878917
- [Result] Anton RF, O'Malley SS, Ciraulo DA, Cisler RA, Couper D, Donovan DM, Gastfriend DR, Hosking JD, Johnson BA, LoCastro JS, Longabaugh R, Mason BJ, Mattson ME, Miller WR, Pettinati HM, Randall CL, Swift R, Weiss RD, Williams LD, Zweben A; COMBINE Study Research Group. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA. 2006 May 3;295(17):2003-17. doi: 10.1001/jama.295.17.2003. PMID 16670409
- [Derived] Acin MT, Rueda JR, Saiz LC, Parent Mathias V, Alzueta N, Sola I, Garjon J, Erviti J. Alcohol intake reduction for controlling hypertension. Cochrane Database Syst Rev. 2020 Sep 21;9(9):CD010022. doi: 10.1002/14651858.CD010022.pub2. PMID 32960976
- [Derived] Falk DE, O'Malley SS, Witkiewitz K, Anton RF, Litten RZ, Slater M, Kranzler HR, Mann KF, Hasin DS, Johnson B, Meulien D, Ryan M, Fertig J; Alcohol Clinical Trials Initiative (ACTIVE) Workgroup. Evaluation of Drinking Risk Levels as Outcomes in Alcohol Pharmacotherapy Trials: A Secondary Analysis of 3 Randomized Clinical Trials. JAMA Psychiatry. 2019 Apr 1;76(4):374-381. doi: 10.1001/jamapsychiatry.2018.3079. PMID 30865232
- [Derived] Zarkin GA, Bray JW, Aldridge A, Mitra D, Mills MJ, Couper DJ, Cisler RA; COMBINE Cost-Effectiveness Research Group. Cost and cost-effectiveness of the COMBINE study in alcohol-dependent patients. Arch Gen Psychiatry. 2008 Oct;65(10):1214-21. doi: 10.1001/archpsyc.65.10.1214. PMID 18838638
- [Derived] Anton RF, Oroszi G, O'Malley S, Couper D, Swift R, Pettinati H, Goldman D. An evaluation of mu-opioid receptor (OPRM1) as a predictor of naltrexone response in the treatment of alcohol dependence: results from the Combined Pharmacotherapies and Behavioral Interventions for Alcohol Dependence (COMBINE) study. Arch Gen Psychiatry. 2008 Feb;65(2):135-44. doi: 10.1001/archpsyc.65.2.135. PMID 18250251